CLINICAL TRIAL: NCT02530788
Title: Perioperative High-dose Selenium Supplementation in Patients With Left Ventricular Assist Device - a Double Blinded Randomised Controlled Trial
Brief Title: High-dose Selenium Supplementation in Patients With Left Ventricular Assist
Acronym: SOS-LVAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: biosyn Arzneimittel GmbH (Industry); Cardiodevice Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-036
Record Dates: First submitted 2015-08-17; First posted 2015-08-21 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Ventricular Dysfunction, Left
Keywords: Heart Failure; Cardiac Surgery; Ventricular Assist Device; Selenium
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure | interventions — Sodium Selenite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selenium Supplement (sodium selenite) (Active Comparator): Active arm receiving Selenium in form of sodium selenite
  Interventions: Drug: Selenium Supplement (sodium selenite)
- Placebo (Placebo Comparator): Placebo arm receiving Sodium Chloride solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selenium Supplement (sodium selenite) — On the evening before operation the patient receives the first dosage of Selenium (300µg orally) orally as a pill.
  After induction of anaesthesia and before being put on the heart-lung-machine the patient receives 3000µg Selenium as sodium selenite (selenase® T) intravenous (as bolus infusion in the space of 30 minutes). In addition the patient gets 1000µg Selenium as sodium selenite (selenase® T) intravenous as bolus infusion in the space of 30 minutes after admission to ICU. On every POD the patient receives 1000µg Selenium as sodium selenite (selenase® T) intravenous as bolus infusion in the space of 30 minutes (until transfer to standard care unit or maximum substitution until 13th POD).
  Other Names: Selenase (R) 300 RP; Selenase (R) T
  Arms: Selenium Supplement (sodium selenite)
Drug: Placebo — On the evening before operation the patient receives the first dosage of placebo orally as a pill.
  After induction of anaesthesia and before being put on the heart-lung-machine the patient receives placebo intravenous (as bolus infusion in the space of 30 minutes). In addition the patient gets placebo intravenous as bolus infusion in the space of 30 minutes after admission to ICU. On every POD the patient receives placebo intravenous as bolus infusion in the space of 30 minutes (until transfer to standard care unit or maximum substitution until 13th POD).
  Arms: Placebo

SUMMARY:
This planned pilot study is a monocentric, prospective, double-blind randomized and placebo controlled clinical study. The SOS-LVAD Trial can be assigned to the clinical Phase III.

The aim of the present trial is to provide the scientific rationale for a large multicenter clinical trial, investigating the effects of perioperative high dose selenium supplementation in high-risk cardiac surgical patients undergoing complicated open heart surgery with prolonged time on cardiopulmonary bypass (CPB) and LVAD Implant. The investigators hypothesize that the therapeutic strategy tested in this randomized trial may contribute to a faster independency from life-sustaining technologies in the ICU and a decrease of postoperative morbidity and mortality. Before proceeding to the large-scale, definitive trial, the investigators propose to conduct a pilot study of the definitive randomized trial, to determine the feasibility of the study protocol.

ELIGIBILITY:
Inclusion criteria:

* Patients with chronic left ventricular heart failure, who undergo LVAD Implant surgery (including other heart surgery)
* Full aged, contractually capable, male and female patients
* Patients that are capable and willing to understand and obey the instructions of the study staff.
* Signed informed consent

Exclusion criteria:

* Selenium intoxication
* Patients with contraindications to the planned intervention, due to diseases
* Severe exacerbation of comorbidities such as renal failure requiring dialysis or liver dysfunction (defined as bilirubin >2mg/dl)
* Known hypersensitivity to the trial medication (selenase® 300 RP, selenase® T), to any of the constituents of the solution or to the placebo
* Patients that are not contractually capable; Patients accommodated to a facility by court order or public authority
* Pregnancy or lactation period
* Women at reproductive age, without suitable contraception
* Patients in a relationship of dependency or in employment with the head of study's
* Underaged
* No signed informed consent
* Simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Composite Outcome: independence from specific ICU procedures | postoperative day 28
  As primary outcome, the investigators have chosen a composite outcome. This allows to assess the postoperative process of the included patients irrespective of extrinsic sources of irritation (e.g. daily routine, clinic based processes). The independency from specific ICU procedures is taken as a primary target (time is taken from postoperative admission to ICU after implantation of LVAD until the end of the characteristic ICU procedures):
  * mechanical ventilation
  * vasopressor therapy
  * mechanical circulatory support
  * renal replacement therapy

SECONDARY OUTCOMES:
Mortality | postoperative day 28
  via telephone enquiry
Persistent organ dysfunction | postoperative day 7
  Persistent organ dysfunction quantified upon day 7 (or upon day of discharge from hospital) with "Sequential Organ Failure Assessment Score" (SOFA), "Multiple Organ Dysfunction Score" (MODS) and "Simplified Acute Physiology Score" (SAPS), daily quantification while ICU stay
Incidence of nosocomial infections acquired at ICU | participants will be followed for the duration of hospital stay, an expected average of 5-10 days
Acute renal failure | participants will be followed for the duration of hospital stay, an expected average of 5-10 days
  (quantified with RIFLE score)
Mechanical Ventilation | participants will be followed for the duration of hospital stay, an expected average of 5-10 days
  Time of mechanical ventilation (measured in hours after successful intubation) and necessity of re-intubation
postoperative delirium | participants will be followed for the duration of hospital stay, an expected average of 5-10 days
  Evaluation of delirium by confusion assessment method: CAM-ICU score
Selenium concentration in whole blood, activity of glutathion-peroxidase, concentration of Selenoprotein-P (Sel-P) | preoperative, by the end of surgery, on day 1, 3, 5, 7, 13, and if the patient is still in hospital, on day 28.
Quality of Life | postoperative day 28
  The patients individual "Quality of Life" (pre- and postoperative) quantified with "MACNEW - Health related quality of life in heart disease - Scale" quantified postoperative upon discharge from hospital and on the 28th POD via telephone inquiry. If the patient cannot be contacted via telephone on the 28th POD, we will try to reach the patient on the following 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Goetzenich, MD, PhD, Principal Investigator — Dep. of Thoracic and Cardiovascular Surgery, University Hospital RWTH Aachen; Christian Stoppe, MD, Principal Investigator — Dep. of Thoracic and Cardiovascular Surgery, University Hospital RWTH Aachen
Locations (1):
- Dep. of Thoracic and Cardiovascular Surgery, University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany